CLINICAL TRIAL: NCT01194986
Title: An Open-label Positron Emission Tomography Study to Evaluate Use of Histamine H3 Receptor Radioligand [11C]AZ12807110 and to Determine Histamine H3 Receptor Occupancy of AZD5213 After Oral Administration to Healthy Volunteers
Brief Title: Evaluation of Histamine H3 Receptor Radioligand [11C]AZ12807110 and Histamine H3 Receptor Occupancy of AZD5213 After Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: D3030C00003; 2009-010702-11 (EudraCT Number)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Brain Distribution of [11C]AZ12807110 and AZD5213
Keywords: Receptor binding; Histamine H3 receptor; binding; radioligand

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilot panel (Experimental): [11C]AZ12807110 distribution and kinetics
  Interventions: Other: [11C]AZ12807110
- Main panel (Experimental): Histamine receptor occupancy reached by AZD5213
  Interventions: Other: [11C]AZ12807110; Drug: AZD5213

INTERVENTIONS:
Other: [11C]AZ12807110 — Radioligand
Drug: AZD5213
  Arms: Main panel

SUMMARY:
The purpose of this study is to investigate features of radioligand [11C]AZ12807110 and how much AZD5213 displaces radioligand from histamine receptors when given together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female volunteers between 20 to 45 years with suitable veins for cannulation or repeated venipuncture (pilot panel)
* Female must be of non-child bearing potential (pilot panel)
* BMI between 18 to 30 30 kg/m2
* Normal MRI scan
* Provision of signed, written and dated informed consent

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of gastrointestinal, hepatic or renal disease
* Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome
* History of severe allergy or hypersensitivity or ongoing allergy or hypersensitivity
* Healthy volunteer suffers from claustrophobia

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Distribution volume (VT) | Venous blood samples for determination of concentrations of AZD5213 in plasma will be taken on many occasions from pre-dose until 48 h post-dose. Single PET measurement will take maximum 2 hours.
Estimation of the plasma concentration resulting in 50% receptor occupancy (Ki, pl). | Venous blood samples for determination of concentrations of AZD5213 in plasma will be taken on many occasions from pre-dose until 48 h post-dose.
  Each healthy volunteer in the main panel will complete 3 PET measurements using radioligand; one at baseline and 2 after treatment with AZD5213.

SECONDARY OUTCOMES:
Adverse events | Collected from Day 1 to follow-up
Vital signs (body temperature, BP and pulse) | Measured at screening, study days -1 to day 3 and at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Björn Paulsson, MD, Study Director — AstraZeneca; Wolfgang Kühn, MD, Principal Investigator — Quintiles AB, Uppsala
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- [Derived] Jucaite A, Takano A, Bostrom E, Jostell KG, Stenkrona P, Halldin C, Segerdahl M, Nyberg S. AZD5213: a novel histamine H3 receptor antagonist permitting high daytime and low nocturnal H3 receptor occupancy, a PET study in human subjects. Int J Neuropsychopharmacol. 2013 Jul;16(6):1231-9. doi: 10.1017/S1461145712001411. Epub 2012 Dec 10. PMID 23217964
- See also: D3030C00003 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1314&filename=D3030C00003_Clinical_Study_Report_Synopsis.pdf